CLINICAL TRIAL: NCT06234267
Title: Eat, Play, Sleep: A Text Message Approach to Promoting Multiple Health Behaviors for Cancer Survivors and Their Informal Caregivers
Brief Title: Eat, Play, Sleep: A Text Message Approach to Promoting Health Behaviors for Cancer Survivors and Their Caregivers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Arizona (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: STUDY00004084
Record Dates: First submitted 2024-01-22; First posted 2024-01-31 (Actual); Last update posted 2025-05-23 (Actual); Status verified 2025-05

CONDITIONS: Cancer Survivors; Neoplasms
MeSH Terms: conditions — Neoplasms | interventions — Eating; Sleep

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Dietary Quality (Experimental): Receive daily text messages for promoting dietary quality.
  Interventions: Behavioral: Eat, Play, Sleep
- Physical Activity (Experimental): Receive daily text messages for promoting physical activity.
  Interventions: Behavioral: Eat, Play, Sleep
- Sleep Hygiene (Experimental): Receive daily text messages for promoting sleep hygiene.
  Interventions: Behavioral: Eat, Play, Sleep

INTERVENTIONS:
Behavioral: Eat, Play, Sleep — The Eat, Play, Sleep study will test health promotion text messages developed following guidelines for text message program development, aligned with established recommendations for diet, physical activity, and sleep in cancer survivorship and prevention. Feasibility of text message delivery and acceptability of the text message content related to dietary quality, physical activity, and sleep hygiene health behaviors will be tested in delivery to participants (cancer survivor/caregiver dyads) who indicate difficulty engaging in dietary quality, physical activity, or sleep hygiene behaviors.

SUMMARY:
Health behavior text message content will be delivered daily over 4-weeks to cancer survivor/caregiver dyads.

ELIGIBILITY:
Inclusion Criteria (survivors and caregivers):

1. ≥18 years old
2. have access to a mobile phone with the ability to receive and send text messages
3. English- or Spanish-speaking
4. free of psychiatric or physical disorders that could interfere with participation (e.g., psychosis, delirium)
5. able to give informed consent in English or Spanish

Survivors must also:

1. have been diagnosed with any solid tumor cancer
2. have completed primary curative treatment at least one month prior to enrollment
3. be able to identify a caregiver to enroll in the study with them
4. report difficulty engaging in dietary quality, physical activity, and/or sleep hygiene behaviors at screening.

Exclusion Criteria:

* Does not meet any of the above criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2024-05-14 (Actual); Primary Completion 2024-11-18 (Actual); Study Completion 2024-12-13 (Actual)

PRIMARY OUTCOMES:
Successful receipt of 95% of text messages sent | 4 weeks
Acceptability of text messages measured by self-report 0-4 likert scale of acceptability of each text message, where 5 is greater acceptability | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Meghan B Skiba, PhD, MS, MPH, RDN, Principal Investigator — University of Arizona
Locations (1):
- University of Arizona Cancer Center, Tucson, Arizona, United States

IPD SHARING:
Plan to Share IPD: No